CLINICAL TRIAL: NCT00418171
Title: An International, Multicenter, Large Simple Trial (LST) To Compare The Cardiovascular Safety Of Ziprasidone And Olanzapine
Brief Title: Large Simple Trial (LST) Of Cardiovascular Safety Of Ziprasidone And Olanzapine- (Zodiac)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281062
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2009-10-26 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone; Olanzapine

INTERVENTIONS:
Drug: Ziprasidone
Drug: Olanzapine

SUMMARY:
The primary objective of the study is to estimate the relative incidence among users of ziprasidone and olanzapine of non-suicide mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly treated for schizophrenia and those receiving continuing treatment will be eligible if the treating psychiatrist is ready to initiate a new antipsychotic medication, and would consider using either ziprasidone or olanzapine as an appropriate therapy.
* Male and female patients who meet all criteria listed below are eligible to be enrolled in this study:
* Diagnosed with schizophrenia
* Willing to provide information on at least one alternate contact person for study staff to contact regarding patient's whereabouts, should the patient be lost-to-follow-up over the course of the study

Exclusion Criteria:

* Progressive fatal disease of a life expectancy which prohibits them from participating in a one year research study
* Previously randomized to study medication and enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18239 (Actual)
Dates: Start 2002-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to estimate the relative incidence among users of ziprasidone and olanzapine of non-suicide mortality within 12 months.

SECONDARY OUTCOMES:
To estimate the relative incidence among users of ziprasidone and olanzapine of all-cause mortality, mortality due to suicide, cardiovascular mortality, mortality due to sudden death | During the year observation period
To estimate the relative incidence among users of ziprasidone and olanzapine of all-cause hospitalization, hospitalization for arrhythmia, myocardial infarction, or diabetic ketoacidosis | During the year observation period
The rate of discontinuation of randomized treatment. | During the year observation period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, ‘Aiea, Hawaii
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Grants Pass, Oregon
  - Pfizer Investigational Site, White Hall, West Virginia

REFERENCES:
- [Derived] Fleischhacker WW, Kane JM, Geier J, Karayal O, Kolluri S, Eng SM, Reynolds RF, Strom BL. Completed and attempted suicides among 18,154 subjects with schizophrenia included in a large simple trial. J Clin Psychiatry. 2014 Mar;75(3):e184-90. doi: 10.4088/JCP.13m08563. PMID 24717389
- [Derived] Kolitsopoulos FM, Strom BL, Faich G, Eng SM, Kane JM, Reynolds RF. Lessons learned in the conduct of a global, large simple trial of treatments indicated for schizophrenia. Contemp Clin Trials. 2013 Mar;34(2):239-47. doi: 10.1016/j.cct.2012.12.001. Epub 2012 Dec 12. PMID 23246610
- [Derived] Strom BL, Eng SM, Faich G, Reynolds RF, D'Agostino RB, Ruskin J, Kane JM. Comparative mortality associated with ziprasidone and olanzapine in real-world use among 18,154 patients with schizophrenia: The Ziprasidone Observational Study of Cardiac Outcomes (ZODIAC). Am J Psychiatry. 2011 Feb;168(2):193-201. doi: 10.1176/appi.ajp.2010.08040484. Epub 2010 Nov 1. PMID 21041245
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281062&StudyName=Large+Simple+Trial+%28LST%29+Of+Cardiovascular+Safety+Of+Ziprasidone+And+Olanzapine%2D+%28Zodiac%29%2E